CLINICAL TRIAL: NCT06434597
Title: A Multicenter, Open, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of SPH5030 Tablets in Subjects With Her2-positive/Mutated Biliary Tract OR Colorectal Cancer.
Brief Title: A Clinical Study of SPH5030 Tablets in the Treatment of Her2-positive/Mutated Biliary Tract OR Colorectal Cancer Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH5030-201
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract or Colorectal Cancer With Her2-positive/Mutated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH5030 (Experimental)
  Interventions: Drug: SPH5030

INTERVENTIONS:
Drug: SPH5030 — SPH5030：Oral, QD, 600mg

SUMMARY:
To evaluate the efficacy and safety of SPH5030 tablets in subjects with Her2-positive/mutated biliary tract OR colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic and/or unresectable advanced colorectal adenocarcinoma, or locally advanced, recurrent, metastatic and/or unresectable advanced biliary tract carcinoma
2. HER2 positive or HER2 gene mutation;
3. Meet the requirements of previous treatment;
4. ECOG performance status of 0 or 1；
5. Expected survival ≥ 3 months;
6. No serious abnormalities in hematopoietic function, liver or kidney function;
7. Females who are not pregnant, non-lactating.. Subjects who complied with the contraceptive requirements of the protocol.;
8. Fully informed subjects who voluntarily sign the ICF.

Exclusion Criteria:

1. Subjects who have previously received anti-HER2 molecular targeted therapy;
2. Subjects who have been treated with any other clinical trial drug within 4 weeks prior to the first dose;
3. Subjects with uncontrolled or severe cardiovascular and cerebrovascular diseases; Subjects with severe lung disease; 4. Subjects who may have conditions that affect the absorption, distribution, metabolism, or excretion of the study drug determined by the investigator;

5 Subjects who are taking potent CYP3A4 or CYP2C8 inhibitors or inducers; 6 Subjects with other malignancies in the past 5 years; 7 Subjects with CNS system metastasis with clinical symptoms; 8 Subjects who do not meet the protocol requirements for hepatitis B and C at screening, have a history of immunodeficiency, or other acquired、congenital immunodeficiency diseases, or have a history of organ transplantation; 9. Other situations that do not meet the requirements of the protolol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.

SECONDARY OUTCOMES:
Duration of remission (DOR) | Approximately 2 years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause.
Disease control rate (DCR) | Approximately 2 years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Progression-free survival (PFS) | Approximately 2 years
  From the start date of study treatment to the date of progression disease or death , whichever occurred first.
Overall Survival (OS) | Approximately 2 years
  Determination of the overall survival times of all patients
Incidence of Treatment-Emergent Adverse Events | Approximately 2 years
  Adverse event type, incidence, duration

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Beijing Friendship Hospital，Capital Medical University, Beijing
  - Chinese PLA General hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Affiliatedf Hospital of AFMU, Beijing
  - XiangYa Hospital CentralSouth University, Changsha
  - Changzhi People's Hospital, Changzhi
  - Fujian Cancer Hospital, Fuzhou
  - General Hospital of Fuzhou, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Hengshui People's Hospital, Hengshui
  - Yunnan Cancer Hospital, Kunming
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai General Hospital, Shanghai
  - The Third Affiliated Hospital of Air Force Medical University, Shanghai
  - Zhongshan Hospital, Shanghai
  - Shantou University Medical College Cancer Hospital, Shantou
  - Liaoning Cancer Hospital, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Medical University Cancer institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Affiliated Hospital of Jiangnan University, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou